CLINICAL TRIAL: NCT06956456
Title: Effects of a 12-week Supervised or Home-based Multicomponent Training Program on Psychological, and Physical Variables in Fibromyalgia Patients
Brief Title: Supervised and Home Training in Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bari Aldo Moro (Other)
Responsible Party: Principal Investigator, Luca Poli, Dr., University of Bari Aldo Moro
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7595
Record Dates: First submitted 2025-04-24; First posted 2025-05-04 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Fibromyalgia
Keywords: mental and physical well-being; anxiety-depressive symptoms; fisical fitness
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Supervised Multicomponent Training (SMCT) (Experimental): subjects assigned to the SMCT group will perform a supervised training protocol defined multicomponent training, which includes aerobic, resistance and flexibility components.
  Interventions: Other: Supervised Multicomponent Training Protocol
- Non-Supervised Home-Based Multicomponent Training (NSMCT) (Experimental): subjects assigned to the NSMCT group will perform a non-supervised home-based training protocol defined multicomponent training, which includes aerobic, resistance and flexibility components.
  Interventions: Other: Non-Supervised Home-Based Multicomponent Training Protocol
- Waiting List Control Group (WLCG) (No Intervention): Subjects assigned to the WLCG group will not engage in any structured physical activity throughout the intervention period, continuing with their usual lifestyle, and will be placed on a waiting list, ensuring their participation in adapted physical activity at the end of the 12-week intervention.

INTERVENTIONS:
Other: Supervised Multicomponent Training Protocol — Supervised Multicomponent Training Protocol
  Each session consists of:
  Warm-up (10 minutes): Low-intensity walking (Borg scale 10-11) to increase heart rate, improve blood flow, and prepare joints.
  Main phase (40 minutes):
  Aerobic exercises: Controlled jumping jacks, step-ups, alternating knee lifts, lateral steps, and leg lifts.
  Mobility exercises: Thoracic extensions, cat-to-cows, overhead stretching with a stick, and hip internal rotations (1-3 sets, 30-60 seconds per exercise).
  Resistance training: Gradual progression of 8 exercises targeting major muscle groups, such as squats, bicep curls, shoulder presses, and rows (1-3 sets, 10-15 reps, RPE 13-15).
  Cool-down (10 minutes): Breathing exercises and stretching (1-3 sets, 10-30 seconds per stretch).
  Arms: Supervised Multicomponent Training (SMCT)
Other: Non-Supervised Home-Based Multicomponent Training Protocol — Participant will receive a personalized exercise plan tailored to their fitness level.
  Each session consists of:
  Warm-up (10 minutes): Low-intensity walking (Borg scale 10-11) to increase heart rate, improve blood flow, and prepare joints.
  Main phase (40 minutes):
  Aerobic exercises: Controlled jumping jacks, step-ups, alternating knee lifts, lateral steps, and leg lifts.
  Mobility exercises: Thoracic extensions, cat-to-cows, overhead stretching with a stick, and hip internal rotations (1-3 sets, 30-60 seconds per exercise).
  Resistance training: Gradual progression of 8 exercises targeting major muscle groups, such as squats, bicep curls, shoulder presses, and rows (1-3 sets, 10-15 reps, RPE 13-15).
  Cool-down (10 minutes): Breathing exercises and stretching (1-3 sets, 10-30 seconds per stretch).
  Arms: Non-Supervised Home-Based Multicomponent Training (NSMCT)

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of supervised multicomponent training (MCT) on physiological parameters, physical fitness, mental well-being, and quality of life in subjects with a history of Fibromyalgia, compared to a non-supervised home-based MCT protocol and a waitlist control group (WLCG). The main questions it aims to answer are:

Does supervised MCT or non-supervised home-based MCT protocol improve physiological parameters, physical fitness, mental well-being, and overall quality of life compared to a waitlist control group (WLCG)? Does supervised MCT provide superior physiological an psychological improvements compared to a non-supervised home-based MCT protocol?

Researchers will compare:

supervised MCT (a combination of aerobic, mobility, and resistance training exercises) and non-supervised home-based MCT protocol to see if these interventions improve fitness, health, psychological and quality of life outcomes compared to WLCG (participants not engaging in structured physical activity during the study), and if there will be significant differences between supervised MCT and non-supervised home-based MCT protocol.

Participants will:

Complete assessments of anthropometric, physical fitness, and psychological parameters at baseline (T0) and after 12 weeks (T1).

Be randomly assigned to one of three groups.

Engage in a 12-week of non-supervised home-based MCT protocol or structured MCT program supervised by exercise professionals, including:

Warm-up sessions (10 minutes, low-intensity walking). Main sessions (40 minutes): aerobic, mobility, resistance (MCT), only-aerobic (AT) exercises.

Cool-down sessions (10 minutes): breathing and stretching exercises.

This study will provide insights into the efficacy of tailored physical activity interventions for Fibromyalgic patients.

ELIGIBILITY:
Inclusion Criteria:

* Women/Men
* Diagnosis of fibromyalgia
* Age between 18 and 75 years at the time of initial treatment;
* Signature of a written informed consent form (or their legally recognized representatives must sign) indicating that the patient understood the purpose and procedures required for the study and is willing to participate in the study;
* Sedentary lifestyle (subjects who have not followed WHO guidelines for aerobic and resistance exercise in the past 3 months);
* Positive medical specialist assessment of noncompetitive physical activity practice

Exclusion Criteria:

* Expected absence for more than one week during the intervention period
* Absence of a medical certificate of suitability for non-competitive sports
* Severe musculoskeletal or joint disorders with significant mobility limitations
* Uncontrolled hypertension or untreated heart disease;
* Pshychiatric disorders;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change in lower body strength | 12-weeks
  30-s chair stand (30CST) test: Sit-to-stand from a chair during 30 seconds (measured in seconds)
Change in functional mobility | 12-weeks
  Timed Up and Go (TUG) Test (measured in seconds)
Change in Handrigp Strength | 12-weeks
  Handgrip Strength (HGS) test: muscle strength measured with manual dynamometers (Kgf)
Change in aerobic capacity | 12-weeks
  2-Minute Step Test (TMST): march in place for 2 minutes, lifting their knees to a height halfway between the iliac crest and the patella.The number of full knee lifts (repetitions) completed in 2 minutes is recorded.
Change in lower body flexibility | 12-weeks
  Chair Sit-and-Reach Test: measures lower body flexibility (hamstrings and lower back) in centimeters (cm). It involves sitting on a chair, extending one leg, and reaching toward the toes to assess mobility. The measurement is taken by recording the distance between the fingertips and the toes. Positive score (+): Fingertips go past the toes.Zero score (0): Fingertips touch the toes. Negative score (-): Fingertips fall short of the toes.
  A ruler or tape measure is used to record the exact distance.
Change in upper body flexibility | 12-weeks
  Back Scratch Test: measures upper body flexibility, particularly shoulder mobility, in centimeters (cm). It involves reaching one hand over the shoulder and the other behind the back to touch or overlap fingers.
  Positive score (+): Fingers overlap (measured as the overlap distance). Zero score (0): Fingers just touch. Negative score (-): Fingers do not touch (measured as the gap distance).
  A ruler or tape measure is used to record the exact distance.
Change in psychological parameters (depression) | 12-weeks
  Beck Depression Inventory (BDI): measures depression severity using a numerical score. It consists of 21 items, each rated on a 4-point scale (0 to 3) based on symptom severity.
  Total score range: 0 to 63 (higher scores indicate more severe depression).
  Interpretation:
  0-13: Minimal depression 14-19: Mild depression 20-28: Moderate depression 29-63: Severe depression
  The final score is obtained by summing the responses.
Change in psychological parameters (anxiety). | 12-weeks
  State-Trait Anxiety Inventory (STAI-Y): measures anxiety levels using a numerical score. It consists of 20 items assessing temporary (state) anxiety on a 4-point scale (1 = not at all to 4 = very much so).
  Total score range: 20 to 80 (higher scores indicate greater anxiety).
  Interpretation:
  20-37: Low anxiety 38-44: Moderate anxiety 45-80: High anxiety
  The final score is obtained by summing the responses.
Change in psychological parameters (enjoyment). | 12-weeks
  he Physical Activity Enjoyment Scale (PACES) is a self-report questionnaire used to measure an individual's enjoyment of physical activity. It assesses positive and negative feelings related to exercise to evaluate motivation and adherence potential.
  It include 18 items rated on a 7-point Likert scale (from 1 = strongly disagree to 7 = strongly agree). Some items are reverse-scored. After adjusting reverse-scored items, all scores are summed to give a total score ranging from 18 to 126, with higher scores indicating greater enjoyment of physical activity.
  A higher total score suggests a more positive emotional response to exercise, which is often linked to better adherence and motivation.
Change in psychological parameters (fear of movement). | 12-weeks
  The TSK is a self-report questionnaire designed to assess fear of movement or re-injury due to physical activity, commonly used in patients with chronic pain.
  Scoring and Interpretation:
  The standard TSK has 17 items, each rated on a 4-point Likert scale (1 = strongly disagree to 4 = strongly agree). Some items are reverse-scored. The total score ranges from 17 to 68, with higher scores indicating greater fear of movement. Scores above 37 often suggest clinically significant kinesiophobia.
Change in psychological parameters (anticipated pain). | 12-weeks
  The PCS is a 13-item self-report questionnaire designed to assess exaggerated negative thoughts and feelings related to actual or anticipated pain. It evaluates three components: rumination, magnification, and helplessness.
  Scoring and Interpretation:
  Each item is rated on a 5-point scale (0 = not at all to 4 = all the time), yielding a total score from 0 to 52. Higher scores indicate greater levels of pain catastrophizing, which are associated with increased pain perception, emotional distress, and poorer treatment outcomes.
Change in psychological parameters (alexithymia). | 12-weeks
  The TAS-20 is a 20-item self-report questionnaire designed to assess alexithymia, a difficulty in identifying and describing emotions. It measures three dimensions: difficulty identifying feelings, difficulty describing feelings, and externally oriented thinking.
  Scoring and Interpretation:
  Each item is rated on a 5-point Likert scale (1 = strongly disagree to 5 = strongly agree). After reverse-scoring appropriate items, the total score ranges from 20 to 100.
  * 51: Non-alexithymic
  52-60: Possible alexithymia
  * 61: Alexithymic Higher scores indicate greater difficulty with emotional awareness and expression.
Change in physical activity levels. | 12-weeks
  The GPAQ is a tool developed by the WHO to assess physical activity levels across three domains: work, transport, and leisure. It captures frequency, duration, and intensity of activity, as well as sedentary behavior.
  Scoring and Interpretation:
  Responses are converted into MET-minutes/week (Metabolic Equivalent Tasks) for each domain. Total physical activity is classified into low, moderate, or high levels based on WHO guidelines. Higher MET scores indicate greater physical activity engagement.
Change in psychological parameters (pain severity). | 12-weeks
  The BPI is a self-report tool used to assess pain severity and the impact of pain on daily functioning. It evaluates both the intensity of pain and how it interferes with aspects of life such as mood, walking, work, and sleep.
  Scoring and Interpretation:
  Pain severity and interference are each rated on 0-10 scales. Scores are averaged separately for severity and interference:
  Severity: 0 = no pain, 10 = worst possible pain.
  Interference: 0 = no interference, 10 = complete interference. Higher scores indicate more severe pain and greater disruption to daily life.
Change in psychological parameters (pain intensity). | 12-weeks
  The NRS is a simple, self-reported tool where individuals rate their current pain intensity on a scale from 0 (no pain) to 10 (worst imaginable pain).
  Scoring and Interpretation:
  Patients select a number that best represents their pain level.
  0: No pain
  1-3: Mild pain
  4-6: Moderate pain
  7-10: Severe pain It's commonly used to monitor pain over time or in response to treatment.
Change in psychological parameters (fatigue). | 12-weeks
  The MAF is a self-report tool designed to assess fatigue across multiple dimensions, including severity, distress, impact on daily activities, and timing, over the past week.
  Scoring and Interpretation:
  The MAF includes 16 items, with most rated on a 10-point scale. It yields a Global Fatigue Index (GFI) ranging from 1 to 50, where higher scores indicate greater fatigue. The GFI provides a comprehensive view of how fatigue affects quality of life.
Change in psychological parameters (sleep quality). | 12-weeks
  The MOS Sleep Scale consists of 12 items assessing sleep quality, disturbances, and patterns, using a 5-point Likert scale. The scores are summed to produce subscale scores for sleep disturbance, sleep adequacy, and sleep problems. Higher scores on the disturbance subscale indicate greater sleep difficulties, while higher scores on the adequacy subscale suggest better sleep quality. Scores are interpreted based on the overall sleep impact, with higher scores reflecting poorer sleep quality.
Change in psychological parameters (psychophysical well-being). | 12-weeks
  The SF-36 consists of 36 items assessing eight health domains: Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role Emotional, and Mental Health. Responses are scored on a 0-100 scale, with higher scores indicating better health status. Domain scores are then combined to create a Physical Component Summary (PCS) and a Mental Component Summary (MCS), which provide an overall measure of physical and mental well-being.
Change in psychological parameters (fibromyalgia impact). | 12-weeks
  The FIQ consists of 21 items, assessing the impact of fibromyalgia on physical functioning, work, pain, fatigue, and sleep. Responses are rated on a scale from 0 to 10, with higher scores indicating greater impairment. The total score ranges from 0 to 100, with higher scores reflecting a greater impact of fibromyalgia on the individual's daily life and well-being.
Cahnge in upper body strength | 12-weeks
  The Arm Curl Test measures upper body strength and endurance, typically performed by having participants repeatedly curl a weighted dumbbell (5 pounds for women, 8 pounds for men) for as many repetitions as possible in 30 seconds.
  Scoring and Interpretation: The score is the total number of successful curls completed within 30 seconds. A higher number of curls indicates better upper body strength and endurance. Scores are interpreted based on age and gender norms, with higher scores reflecting better physical fitness.
Change in body mass index | 12-weeks
  BMI is calculated by dividing a person's weight in kilograms by their height in meters squared (kg/m²).
  Underweight: BMI < 18.5
  Normal weight: BMI 18.5-24.9
  Overweight: BMI 25-29.9
  Obesity: BMI ≥ 30
  A higher BMI typically indicates an increased risk for health issues related to weight, while a lower BMI may signal malnutrition or underweight.

CONTACTS AND LOCATIONS:
Overall Officials: Luca Poli, Dr., Principal Investigator — University of Bari Aldo Moro
Locations (1):
- Società Ginnastica Angiulli, Bari, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-04-24): https://cdn.clinicaltrials.gov/large-docs/56/NCT06956456/Prot_SAP_000.pdf
  • Informed Consent Form (2025-04-24): https://cdn.clinicaltrials.gov/large-docs/56/NCT06956456/ICF_001.pdf